CLINICAL TRIAL: NCT03823469
Title: Evaluating the Impact of a Culinary Coaching Telemedicine Program on Body Weight and Metabolic Outcomes - A Randomized Controlled Trial
Brief Title: Evaluating the Impact of a Culinary Coaching Tele-medicine Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Ran Polak, CHEF Coaching program director, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P002115
Record Dates: First submitted 2019-01-15; First posted 2019-01-30 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Overweight; Obesity
Keywords: Home cooking; Telemedicine; Nutrition; Health coaching
MeSH Terms: conditions — Overweight; Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Nutritional counseling + CCTP (Active Comparator): Nutritional counseling + Culinary Coaching Telemedicine Program (CCTP)
  Interventions: Behavioral: CCTP; Behavioral: Nutritional counseling
- Control: Nutritional counseling only (Active Comparator): Two 30-minute nutritional counseling sessions
  Interventions: Behavioral: Nutritional counseling

INTERVENTIONS:
Behavioral: CCTP — Twelve weekly one-on-one 30-minute tele-sessions through video conference. At the first session, subjects identify their vision regarding home cooking and 3-month goals. During each subsequent meeting, subjects will review their progress towards reaching the prior week's culinary goals and identify goals for the coming week, using a self-discovery process. When patients detect a new culinary skill that is necessary for their progress, s/he will either be taught through discussions or referred to active learning from a Culinary Resource Center.
  Arms: Intervention: Nutritional counseling + CCTP
Behavioral: Nutritional counseling — Two 30-minute nutritional counseling sessions

SUMMARY:
Introduction: Obesity is a major public health problem and adopting healthy lifestyle habits, while effective, is challenging in real-world settings. Culinary coaching is a behavioral intervention that aims to improve nutrition and overall health by facilitating home cooking through an active learning process that combines culinary training and health coaching. Our goal is to evaluate whether a culinary coaching telemedicine program (twelve 30-minute sessions) will significantly improve outcomes among subjects with overweight or obesity.

General hypothesis: A culinary coaching telemedicine program will result in significant weight loss, and improvement in culinary attitude and self-efficacy, nutritional intake, and metabolic outcomes.

Methods: This is a two-site, 36-month randomized controlled trial in which study participants between the ages of 25 to 70, with 27.5 ≤ BMI ≤ 35 Kg/m2 will be randomly assigned to nutritional counseling combined with a structured culinary coaching program or to nutritional counseling group (18 intervention, 18 control at each site). Intervention will include a 3-month culinary coaching telemedicine program with outcome data collected periodically for 12 months. The pre-defined primary outcome is body weight loss at 6 months, and secondary outcomes include change in body weight and composition at 1 year, as well as culinary attitudes and self-efficacy through a validated questionnaire, nutritional intake, lipid profile, blood pressure, and HgA1c (glycated hemoglobin); and participants' perception of the program.

Potential impact: The investigators believe that this program has a potential to be a viable tool in promoting effective and scalable home cooking interventions aimed at improved nutrition and health outcomes in overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Stable oral medications for the past 3 months (or with type 2 diabetes mellitus who are well controlled (Hga1C<7.5) and on stable oral medications for the past 6 months
* Body mass index (BMI) equal or greater than 27.5 Kg/m2 and equal or lower than 35 Kg/m2.
* Subjects who will agree to be randomized to either one of the 2 study arms
* Accessible by phone, and able to watch online videos.
* English (Spaulding) or Hebrew (Sheba) speaking subjects
* At least self-report one visit with a physician or dietitian in the last 12 months.

Exclusion Criteria:

* Pregnant or nursing women within the past 6 months
* Weight loss medications (e.g., topiramate, buproprion, orlistat) within the past 6 months or medications likely to cause weight gain or prevent weight loss (e.g., corticosteroids, lithium, olanzapine, risperidone, clozapine
* Either type 1 or 2 diabetes who are on insulin
* Uncontrolled hypothyroidism or hyperthyroidism
* Serious medical conditions likely to hinder accurate measurement of weight, or for which weight loss is contraindicated, or which would cause weight loss (e.g., end stage renal disease on dialysis, cancer diagnosis or treatment within 2 years)
* Unstable angina or with myocardial infarction, stroke or atherosclerotic cardiovascular disease procedure within 6 months prior to screening
* Self-reported average consumption of > 14 alcoholic drink per week
* Prior or planned bariatric surgery
* Unintentional weight loss within 6 months of enrollment (≥ 5% of body weight), or Intentional weight loss within 6 months (≥ 5% of body weight)
* Subjects following specific dietetic recommendations (e.g., celiac sprue, cystic fibrosis)
* Subjects with eating disorders, or any psychiatric hospitalization in last year prior to screening.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Body weight at 6 months | Six months
  5% decrease in body weight (kg) in the intervention arm as compared to control. measured by a registered dietitian.

SECONDARY OUTCOMES:
Body weight | Body weight will be obtained at baseline, after the intervention (at 3 months), 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  Body weight (kg), measured by a registered dietitian
Culinary attitude & self-efficacy | Culinary attitude & self-efficacy will be obtained at baseline, after the intervention (at 3 months), 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  Culinary attitudes and self-efficacy will be evaluated by the Cooking With a Chef (CWC) Instrument. This is a 22-item self-administered Likert scale questionnaire that generates three subscales: 1) the cooking techniques and meal preparation self-efficacy subscale (14 items; 1 - not al all confident; 5- extremely confident; sub-scale range 14-70), 2) the negative cooking attitudes subscale (4 items; 1 - strongly disagree; 5 - strongly agree; sub-scale range 4-20), and, 3) the self-efficacy to consume fruit and vegetables subscale (5 items; 1 - not al all confident; 5- extremely confident; sub-scale range 5-25).
Nutritional intake | Nutritional intake will be obtained at baseline, after the intervention (at 3 months), 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  Nutritional intake will be evaluated by a 4-day food record. Intake will be analyzed for its caloric content (kcal), saturated fats(g), trans fats(g), legumes (g), fruits (g), red and processed meat (g), sugars(g), processed food(g), vegetables(g), soft drinks(g), fish(g), whole grain(g), refined grain(g), and monounsaturated fat-saturated fat ratio. Vegetables, legumes, fruits, nuts, whole grains, fish, monounsaturated fat-saturated fat ratio, alcohol, and meat will be aggregate to report Mediterranean index in points (1-9))
Adherence to Mediterranean Diet | Nutritional intake will be obtained at baseline, after the intervention (at 3 months), 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  Adherence to Mediterranean Diet will be evaluated by the validated 14 items Questionnaire of Mediterranean Diet Adherence, extracted by a dietitian from a 4-day food record (0 - low adherence; 14 - high adherence)
Consumption of ultra-processed | Nutritional intake will be obtained at baseline, after the intervention (at 3 months), 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  Consumption of ultra-processed food will be evaluated by the NOVE food classification, extracted by a dietitian from a 4-day food record (unprocessed or minimally processed foods (g), processed culinary ingredients (g), processed foods (g), ultra processed foods (g))
Blood pressure | Blood pressure will be obtained at baseline, after the intervention (at 3 months), 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  blood pressure (both systolic and diastolic), measured in a seated position by a nurse using a sphygmometer
Lipid profile | Lipid profile will be obtained at baseline, after the intervention (at 3 months), 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  Lipid profile (total cholesterol, HDL-cholesterol, LDL-cholesterol, non-HDL cholesterol and triglycerides), measured from a blood sample drawn
HbA1c | HbA1c will be obtained at baseline, after the intervention (at 3 months), 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  HbA1c, measured from a blood sample drawn
Lean body mass | Lean body mass will be obtained at baseline, and at 6 months after the beginning of the intervention
  Lean body mass (g) will measured using Bone Densitometry
Total fat mass | Total fat mass will be obtained at baseline, and at 6 months after the beginning of the intervention
  Total fat mass (g, %fat) will measured using Bone Densitometry
Trunk fat mass | Trunk fat mass will be obtained at baseline, and at 6 months after the beginning of the intervention
  Trunk fat mass (g, %fat) will measured using Bone Densitometry
Fat distribution | Body composition will be obtained at baseline, and at 6 months after the beginning of the intervention
  Fat distribution will measured using Bone Densitometry. Measurements includes: android fat mass (g, %fat) and gynoid fat mass (g, %fat). Fat distribution will be extracted from Android/ Gynoid
Stages of change in relation to home cooking | Stages of change will be obtained at baseline, after the intervention (at 3 months), 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  Stages of change in relation to home cooking as assessed by the validated University of Rod Island Change Assessment (URICA) Scale. This is a 32-item self-administered Likert scale questionnaire (1 - strongly disagree; 5 - strongly agree). Minimum score - 32, maximum score - 160
Perceived Stress | Perceived stress will be obtained at baseline, after the intervention (at 3 months), 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  Perceived Stress, evaluated by the validated Perceived Stress Scale. This is a 10-item self-administered Likert scale questionnaire (0 - never; 4 - very often). Minimum score - 0, maximum score - 10.
Subject perceptions of the program | subjects perception of the program will be obtained using open ended questionnaires at baseline, 6 months after the beginning of the intervention, and 12 months after the beginning of the intervention
  Information about subjects' experiences (e.g., feelings during the CCTP; difficulties, dilemmas, and challenges during the program) will be evaluated using a structured open-ended questionnaire.
Subject perceptions of the program | Subjects perception of the program will be obtained using in-depth interview after the intervention (at 3 months).
  Information about subjects' experiences (e.g., feelings during the CCTP; difficulties, dilemmas, and challenges during the program) will be evaluated using In-depth semi-structured interview.
Coping with Stress | Coping with stress will be obtain through the 2 months of the pick COVID-19 epidemic
  Overall resiliency to cope with the COVID-19 epidemic with be obtained through the Brief Resilient Coping Scale and copying strategies through the Brief Cope scale

CONTACTS AND LOCATIONS:
Overall Officials: Rani Polak, MA, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (2):
- Spaulding Rehabilitation hospitle, Charlestown, Massachusetts, United States
- Sheba Medical Center, Ramat Gan, Israel